CLINICAL TRIAL: NCT04056182
Title: Lofexidine for Management of Opioid Withdrawal With XR-NTX Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: USWM, LLC (dba US WorldMeds) (Industry)
Responsible Party: Principal Investigator, Frances R Levin, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7812
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Opioid-use Disorder
Keywords: opioid use disorder; lofexidine; naltrexon-xr
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lofexidine

STUDY DESIGN:
Intervention Model Description: open label treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lofexidine (Experimental): Lofexidine prescribed as three 0.18mg tablets taken orally 4 times daily at 4-to 6-hour intervals for 2-10 days for the management of opioid withdrawal symptoms prior to receiving Vivitrol.
  Interventions: Drug: Lofexidine 0.18 MG

INTERVENTIONS:
Drug: Lofexidine 0.18 MG — Lofexidine prescribed as three 0.18mg tablets taken orally 4 times daily at 4-to 6-hour intervals for 2-10 days for the management of opioid withdrawal symptoms prior to receiving Vivitrol.
  Other Names: Lucemyra

SUMMARY:
This is an open-label pilot trial to evaluate the safety and tolerability of lofexidine in the management of opioid withdrawal symptoms while initiating outpatient treatment with naltrexone. The initiation procedure will be a flexible detoxification lasting 2 to 10 days concluding with the injection of XR-Naltrexone (Vivitrol). Vivitrol is a long-acting injection that contains enough medicine to last for one month blocking the effects of opioids.

DETAILED DESCRIPTION:
This is an open-label pilot trial to evaluate the safety and tolerability of lofexidine in the management of opioid withdrawal symptoms while initiating outpatient treatment with naltrexone. Lofexidine is a nonopioid prescription medicine used in adults to help with the symptoms of opioid withdrawal that may happen when a person stops taking an opioid suddenly. The initiation procedure will be a flexible detoxification lasting 2 to 10 days concluding with the injection of XR-Naltrexone (Vivitrol). Vivitrol is a long-acting injection that contains enough medicine to last for one month blocking the effects of opioids. Lofexidine will be fixed-flexible dosing started on day 1 with maximum dose being three 0.18mg tablets taken orally 4 times daily at 4-to 6-hour intervals. Lofexidine treatment will continue throughout the detoxification, up to 10 days, and will be discontinued with a gradual dose reduction over 2 to 4 days. Precipitated withdrawal symptoms are treated with lofexidine, clonazepam, and other comfort medications. After the induction patients will be seen at the clinic for 8 weeks. Twice weekly for the first month and weekly for weeks 5-8. A second Vivitrol injection will be provided at week 4.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-60
* Meets DSM-5 criteria of current opioid use disorder present for at least six months, supported by a positive urine for opioids on day of consent
* Seeking treatment for opioid use disorder
* Capable of giving informed consent and complying with study procedures
* History of opioid withdrawal

Exclusion Criteria:

* Meets DSM-5 criteria for substance use disorder other than opioid as the primary diagnosis
* Having a comorbid psychiatric diagnosis that might interfere with participation or make participation hazardous, such as an active psychotic disorder or current suicide risk
* Methadone maintenance or long-acting agonist (buprenorphine) treatment -Buprenorphine maintenance treatment
* Known history of allergy, intolerance, or hypersensitivity to candidate medication
* Pregnancy, lactation, or failure to use adequate contraceptive methods in female patients
* Unstable medical conditions, which might make participation hazardous such as uncontrolled hypertension (blood pressure >150/100), acute hepatitis, uncontrolled diabetes, or elevated liver function tests (AST and ALT >3 times the upper limit of normal)
* Legally mandated to substance use disorder treatment
* Currently physiological dependence on alcohol or sedative-hypnotics that would require a medically supervised detoxification-other substance use diagnoses are not exclusionary
* Painful medical condition that requires ongoing opioid analgesia or anticipated surgery necessitating opioid medications (Clinical interview; psychiatrist)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: FRANCES R (MD) R LEVIN, MD, Principal Investigator — New York Psychiatric Institute
Locations (1):
- STARS/NYSPI-Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lofexidine
Started | 20
Completed | 3
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Lofexidine
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants] — sex based on self report
  Participants
    Female | 4
    Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 1
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Successful Vivitrol Induction
Description: number of participants inducted onto Vivitrol
Time Frame: up to 10 days of detoxification and induction
Population: number of individuals who enrolled in the trial and initiated the detoxification/induction process
Measure: Count of Participants; unit: Participants
Arm/Group | Lofexidine
Number analyzed (Participants) | 20
Participants | 10

ADVERSE EVENTS:
Time Frame: 2-10 day induction period followed by 8 weeks of the trial
Arm/Group | Lofexidine
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lofexidine (N=20)
inpatient detoxification (General disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lofexidine (N=20)
dizziness (General disorders) | 12 (12)
diarrhea (Gastrointestinal disorders) | 4 (4)
insomnia (General disorders) | 4 (4)
anxiety (Psychiatric disorders) | 2 (2)
depression (Psychiatric disorders) | 2 (2)
fatigue (General disorders) | 2 (2)
GI upset (Gastrointestinal disorders) | 2 (2)
headache (General disorders) | 2 (2)
orthostasis (Cardiac disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2)
anhedonia (General disorders) | 1 (1)
blurred vision (Eye disorders) | 1 (1)
drowsiness (General disorders) | 1 (1)
hyporexia (Gastrointestinal disorders) | 1 (1)
hypotension (Cardiac disorders) | 1 (1)
muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
weight loss (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT04056182/Prot_SAP_000.pdf